CLINICAL TRIAL: NCT06173674
Title: The Feasibility and Acceptability of a Music Intervention to Reduce Preoperative Anxiety (Fa-MIPA Study) in Older Patients Undergoing Cardiac Surgery or Transcatheter Aortic Valve Implantation (TAVI) Procedure
Brief Title: The Feasibility and Acceptability of a Music Intervention to Reduce Preoperative Anxiety in Older Patients
Acronym: fa-MIPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, prof. dr. Koen Milisen, Full professor, KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S68344
Record Dates: First submitted 2023-11-20; First posted 2023-12-18 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Preoperative Care; Preoperative Anxiety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music intervention (Experimental): The music intervention will consist of three components, including 1) playlist composition, 2) music intervention delivery, and 3) cleaning or disinfection of the equipment.
  Interventions: Other: Music intervention

INTERVENTIONS:
Other: Music intervention — The music intervention will consist of three components including:
  1. Playlist composition Six music genres playlists will be offered to patients, including Classical Music, Country Music, Folk Music, Hymns and Reglious Music, Jazz and Swing Music, Popular/Easy Listening/RNB and Soundtrack Music. Patients can also add their favourite music to the list as well.
  2. Music Intervention Delivery The general criteria for intervention delivery are:1) Each session lasts at least 20 minutes; 2) The music will be delivered by a comfortable, wireless, on/off switch noise-cancelling headphone; 3) The volume will be adjusted according to the patient's preference and controlled at 65dB or lower; 4) The order of music in the playlists will be decided by the patient; 5) Music will be delivered in inpatient room and/or waiting area before surgery/procedure.
  3. Cleaning and infection of the equipment We will comply with guidelines on disinfection of materials in the hospital.

SUMMARY:
The goal of this clinical feasibility study is to learn about the acceptability and feasibility of a music intervention in older patients undergoing cardiac surgery and Transcatheter Aortic Valve Implantation (TAVI) procedure.

The primary question it aims to answer is:

• What is the feasibility and acceptability of a music intervention to reduce PA in older patients undergoing cardiac surgery and TAVI?

The secondary question is:

• What is the effect of a music intervention on PA levels and the incidence of POD in older patients undergoing cardiac surgery and TAVI?

Participants will

* listen to music before the surgery/TAVI procedure
* be evaluated for preoperative anxiety levels and postoperative delirium
* be interviewed to learn about their perspectives regarding the music intervention

DETAILED DESCRIPTION:
Background: High levels of preoperative anxiety (PA) have been associated with several complications, including hemodynamic instability, increased intraoperative requirements for anaesthetics, increased risk of postoperative pain, and in some studies an increased incidence of postoperative delirium (POD). Especially for people with reduced physiological reserves such as older patients, PA can independently heighten the risk of mortality or major morbidity. Music intervention stands out as an effective and practical non-pharmacologic intervention on reducing PA levels. Current evidence has proven the effectiveness of music interventions in reducing preoperative anxiety levels; however, the patients' attitudes, preferences, and overall experience of receiving music intervention before surgery are insufficiently explored. Consequently, the investigation of the acceptability of a music intervention among older patients waiting for surgery or other medical procedures is important, as acceptability has emerged as a pivotal factor in the development, assessment, and implementation of a healthcare intervention. Furthermore, it is essential to assess the feasibility of implementing music intervention within the target population, thereby enhancing the overall acceptability of this intervention.

Objectives: The primary objective is to assess the feasibility and acceptability of a music intervention in reducing PA in older patients undergoing cardiac surgery and Transcatheter Aortic Valve Implantation (TAVI) procedure. The secondary objective is to test the effect of the music intervention on preoperative anxiety reduction and the incidence of POD in the target population. Moreover, this study will provide reference for the design of a future randomized controlled trial investigating the relationship between PA and POD in older cardiac surgical patients.

Setting: This feasibility study will be conducted in the Department of Cardiology and Department of Cardiovascular Surgery of the University Hospitals Leuven.

Overall methodology: All potential patients will be identified from the list of patients scheduled for surgery or procedure, and they will be assessed for eligibility after agreeing to participate in this study. They will be provided with an information leaflet with the purpose, process, and potential benefits and harms of this study, as well as the commitment to confidentiality and freedom to withdraw at any time without any consequence. Only the patients willing to participate in the study will be further evaluated to determine their adherence to the inclusion/exclusion criteria. For the eligible patients, we will perform the baseline assessment immediately after obtaining written informed consent from patients.

After admission to hospital, patients will receive music intervention before or during surgery/procedure and perioperative routine postoperative care until discharge. We will assess the preoperative anxiety levels of the patient using validated questionnaires at the baseline and after the music intervention, as well as their perspectives regarding the acceptability and feasibility of music intervention via short interview. Any adverse outcomes related to surgery/procedure or music interventions will also be collected.

In light of feasibility nature of our study, a power calculation is deemed unnecessary, and a sufficient sample size of 30-50, accounting for a 20% attrition rate due to short stays before surgery, leads to a planned minimum recruitment of 70 patients. Four trained study nurses will collect the data under the supervision of PhD student and the promotors. All the data will be firstly collected manually by study nurses, and then will be entered and maintained in the Research Electronic Data Capture (REDCap) database.

Descriptive statistics of demographical information, clinical data, and feasibility and acceptability data will be analysed using suitable numerical and graphical summaries for quantitative data. Paired Samples T-Test will be used for preoperative anxiety level changes before and after the music intervention. The difference of incidence of POD between the group with PA reduction and group without PA reduction will be tested using Chi-squared test. The qualitative data will be analyzed using thematic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients being 60 years or older, scheduled for elective cardiac surgery and Transcatheter Aortic Valve Implantation (TAVI);
* being capable and willing to participate in the study.

Exclusion Criteria:

* cannot use headphones;
* have a history of music-induced seizures;
* have deafness or severe ear diseases such as acute otitis media, eardrum rupture, tinnitus, ear infections, etc.;
* admitted on the day of cardiac surgery;
* have an expected hospital stay of less than 24 hours or a planned intensive care unit stay postoperatively for longer than one day;
* have severe postoperative complications and are unable to be interviewed;
* are currently diagnosed with major psychiatric disease (such as, major depression, generalized anxiety disorder) and dementia as identified in the history of patients file;
* have pre-operative delirium

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Reach | Recruitment, on average of 1 day
  The number and proportion of individuals willing to participate will be calculated, and reasons for refusing will be documented.
Compliance rate | from admission to time just before surgery, on average of 2 days
  The compliance rate refers to one session with 20 minutes or more of music intervention on the day before and on the day of surgery/TAVI procedure.
Acceptability of music intervention | After surgery to discharge, on average of 5 days
  Patients perspective regarding their satisfaction and experience of the music intervention will be asked via a short interview (e.g., Overall, were you satisfied with the music listening before your surgery/procedure? Would you like to listen to music again in a future surgery/procedure?)
Patients' preference of music intervention | After surgery to discharge, on average of 5 days
  Patients' preference regarding intervention details including music selection, number of sessions, duration, setting, and implementation time, will be asked via a short interview (e.g., Do you think listening to music 2 times before surgery is enough to reduce anxiety about the surgery/ procedure? When would you prefer to listen to the music?).
Barriers of receiving music intervention | After surgery to discharge, on average of 5 days
  Barriers of receiving music intervention will be also asked (e.g., Did you experience any problems while listening to music?).

SECONDARY OUTCOMES:
Preoperative anxiety levels (APAIS-A) | from admission to the day of surgery, on average of 2 days
  The preoperative anxiety level will be assessed using the anxiety subscale of Amsterdam Preoperative Anxiety and Information Scale (APAIS-A) before and after receiving the music intervention. APAIS-A consists of 4 items, each of which could be scored from 1 to 5. The score of the APAIS-A is the sum of these four questions, with a scoring range from 4 (not anxious) to 20 (highly anxious).
Preoperative anxiety levels (STAI-6) | from admission to the day of surgery, on average of 2 days
  The preoperative anxiety level will be assessed using six-item Dutch version of the state scale of the Spielberger State-Trait Anxiety Inventory (STAI-6) before and after receiving the music intervention. STAI-6 consists of 6 items, each of which could be scored from 1 (not at all) to 4 (very much so). The sum score varies between 6 and 24, with higher scores indicating higher levels of anxiety.
Preoperative anxiety levels (VAS-A) | from admission to the day of surgery, on average of 2 days
  The preoperative anxiety level will be assessed using VAS-A (Visual Analogue Scale for anxiety) before and after receiving the music intervention. The VAS-A consists of a line which is 10 centimeters in length. Patients are asked to mark a cross on the line based on how they feel during a specified moment in time. A mark at the extreme left end indicates that one feeling not at all anxious. A mark at the extreme right end would indicate that you are feeling the most anxious you could ever imagine.
Preoperative anxiety levels (short interview) | After surgery to discharge, on average of 5 days
  We will also ask patients a few questions regarding their changes in overall status and negative thoughts specific to surgery after receiving the music intervention (e.g., Did you feel more relaxed after listening to music before the surgery/procedure?).
Incidence of postoperative delirium | After surgery to discharge, on average of 5 days
  The incidence of postoperative delirium during all postoperative days will be assessed using 3D-CAM (3-Minute Diagnostic Interview for Confusion Assessment Method) and checking patients' records for the results of the Delirium Observations Scale performed by the nurses on the ward. Medical records will also be retrospectively reviewed using CHART-DEL (Chart-based Delirium Identification Instrument) to identify postoperative delirium.

CONTACTS AND LOCATIONS:
Overall Officials: Koen Milisen, PhD, Principal Investigator — Department of Public Health and Primary Care, Academic Centre for Nursing and Midwifery, KU Leuven
Locations (1):
- University Hospital Leuven, Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analyzed during the current study are available from the corresponding author on reasonable request. As far as requests are in line with the scope and research objectives of the fa-MIPA study.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: On reasonable request
Access Criteria: The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request. As far as requests are in line with the scope and research objectives of the fa-MIPA study.

REFERENCES:
- [Background] Yang KL, Detroyer E, Van Grootven B, Tuand K, Zhao DN, Rex S, Milisen K. Association between preoperative anxiety and postoperative delirium in older patients: a systematic review and meta-analysis. BMC Geriatr. 2023 Mar 30;23(1):198. doi: 10.1186/s12877-023-03923-0. PMID 36997928
- [Background] Stamenkovic DM, Rancic NK, Latas MB, Neskovic V, Rondovic GM, Wu JD, Cattano D. Preoperative anxiety and implications on postoperative recovery: what can we do to change our history. Minerva Anestesiol. 2018 Nov;84(11):1307-1317. doi: 10.23736/S0375-9393.18.12520-X. Epub 2018 Apr 5. PMID 29624026
- [Background] Williams JB, Alexander KP, Morin JF, Langlois Y, Noiseux N, Perrault LP, Smolderen K, Arnold SV, Eisenberg MJ, Pilote L, Monette J, Bergman H, Smith PK, Afilalo J. Preoperative anxiety as a predictor of mortality and major morbidity in patients aged >70 years undergoing cardiac surgery. Am J Cardiol. 2013 Jan 1;111(1):137-42. doi: 10.1016/j.amjcard.2012.08.060. PMID 23245838
- [Background] Wang R, Huang X, Wang Y, Akbari M. Non-pharmacologic Approaches in Preoperative Anxiety, a Comprehensive Review. Front Public Health. 2022 Apr 11;10:854673. doi: 10.3389/fpubh.2022.854673. eCollection 2022. PMID 35480569
- [Background] Aguero-Millan B, Abajas-Bustillo R, Ortego-Mate C. Efficacy of nonpharmacologic interventions in preoperative anxiety: A systematic review of systematic reviews. J Clin Nurs. 2023 Sep;32(17-18):6229-6242. doi: 10.1111/jocn.16755. Epub 2023 May 6. PMID 37149743
- [Background] Bradt J, Dileo C, Shim M. Music interventions for preoperative anxiety. Cochrane Database Syst Rev. 2013 Jun 6;2013(6):CD006908. doi: 10.1002/14651858.CD006908.pub2. PMID 23740695